CLINICAL TRIAL: NCT06283043
Title: Effect of Motor Function, Depression and Sleep Quality on Attention in Parkinson's Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Assoc.Prof., Inonu University
Other Study IDs: 2022/3749
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Movement Disorders (Incl Parkinsonism); Parkinsonian Disorders; Attention Impaired; Movement Disorders, Functional
Keywords: Parkinson; Attention; motor function; sleep
MeSH Terms: conditions — Movement Disorders; Parkinsonian Disorders; Conversion Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: Parkinson's patients will be included and the evaluations specified in the method section will be applied.
- control group: The healthy group will be included and the evaluations specified in the method section will be applied.

SUMMARY:
Our study was planned to analyze motor function, endurance and sleep attention information in Parkinson's patients with detailed and objective measurements.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a neurodegenerative disease that occurs with the loss of dopaminergic neurons in the basal ganglia (BG) and subsequently affects multiple brain regions. There are studies that evaluate executive functions rather than cognitive functions in Parkinson's patients. However, objective evaluations of the attention parameter are quite rare. Accordingly, our study was planned to examine the effects of motor function, depression and sleep on attention in Parkinson's patients with detailed and objective measurements. Parkinson's patients (n=27) and healthy controls (n=27) aged between 40-85 will be included in the study. Balance evaluation of the individuals participating in the study was carried out by functional reaching test, one-leg standing test and Berg balance scale; Endurance with a 30-second sit-and-stand test; reaction time; with mobile application; muscle strength by hand dynamometer; functional mobility with time up and go test; walking speed, with 10 m walk test; attention with the P300 device; depression, with the Beck depression scale; Sleep quality will be assessed with the Pittsburg sleep questionnaire. At the end of the study, the effects of motor functions, sleep and depression on attention will be examined and compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Being 1,2 or 3 according to the Hoehn and yahr scale
* Being between the ages of 40-85
* Being diagnosed with Parkinson's according to UPDS
* Being able to read and write
* Being able to walk independently
* Agreeing to participate in the study after providing detailed information about the research.
* Mini mental test>24

Exclusion Criteria:

* Having severe hearing/visual impairment-loss
* Having an orthopedic, neurological or metabolic disease that may interfere with working
* Having deep brain stimulation applied
* Those with advanced cognitive impairment
* Individuals with dementia
* Patients taking anticholinergic, antidepressive or anxiolytic medications that may affect cognition, and those with other medical or neurological causes that may cause cognitive effects.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parkinson Diseases and Healty Control
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-05 (Estimated)

PRIMARY OUTCOMES:
TUG | second, day 1, Values over 12 seconds indicate the risk of falling
  functional mobility
10 m walking test | second, day 1, lower results indicate better values, higher results indicate worse results
  walking speed
30 sec sit-stand test | again,day 1, higher results indicate better values, lower results indicate worse results
  endurance
berg balance test | score, day 1, The score is between 0-56. A high total score indicates a good result
  balance
one leg stance test | second, day 1, higher results indicate better values, lower results indicate worse results
  balance
functional reach test | centimeter, day 1, higher results indicate better values, lower results indicate worse results
  balance
hand dinamometer | kilogram, day 1, higher results indicate better values, lower results indicate worse results
  strenght
mobil application | second, day 1, lower results indicate better values, higher results indicate worse results
  reaction time
Pittsburg Sleep Quality İndex | score, day 1, The score is between 0-21. A high total score indicates a bad result.
  sleep
Beck Depression | score,day 1, The total score is between 0-63. A high total score indicates that the result is bad.
  depression
P300 | second, day 1, lower results indicate better values, higher results indicate worse results
  attention

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Battalgazi, Turkey (Türkiye)